CLINICAL TRIAL: NCT03355222
Title: Using Eggshell Calcium to Mitigate Fluorosis in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Hawassa University (Other)
Responsible Party: Principal Investigator, Susan Whiting, Professor of Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HU-UoS-EGGSHELL-FLUORIDE
Record Dates: First submitted 2017-11-09; First posted 2017-11-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Fluoride Poisoning; Hemoglobin; Underweight; Stunting; Development; Delayed, Mental; Fluorosis, Dental; Fluorosis; Skeletal; Zinc Deficiency
Keywords: complementary feeding; calcium
MeSH Terms: conditions — Fluoride Poisoning; Thinness; Growth Disorders; Fluorosis, Dental

STUDY DESIGN:
Intervention Model Description: Subjects to be drawn from two simlar villages: one is intervention village and other is control village.
Masking Description: Chickens are how we intervene and this is not possible to "blind'. Two villages will be far apart. We will not disclose nature of intervention to examiners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): No intervention: The community receives no chickens and no special education is provided.
- Experimental: providing chickens and egg shell (Experimental): Experimental: Two chickens are given to each family so that eggs are available for children and of eggshell powder for mothers.
  The community receives these chickens so each designated family has an egg to give to young child. In a subgroup the mother will receive ESP (1000 mg calcium). The community receives information on using egg and has help on caring for chickens.
  Interventions: Behavioral: Promotion of chicken eggs

INTERVENTIONS:
Behavioral: Promotion of chicken eggs — Community is provided with chickens and young children are to receive one egg a day; selected mothers will consume eggshell.
  Arms: Experimental: providing chickens and egg shell

SUMMARY:
Mothers and young children in rural Ethiopia lack sufficient nutrition, and a compounding factor is presence of high levels of fluoride (> 5-10 mg/day) affecting body functions. Interventions involving chickens to provide eggs and eggshell (a source of calcium) are one solution. The overall purpose is to examine how increasing dietary calcium by using eggshell powder (ESP) reduces fluoride (F) absorption in women. It is known calcium binds F to prevent its absorption but application of this to a community based study has not been tested. The aim is to provide chickens to produce eggs for young children and to provide ESP to women (mothers). For children, an egg a day should improve growth and nutritional status. For women, the ESP provides calcium to reduce fluorosis and therefore improve function without affecting iron and zinc status. For the women, blood samples will be tested in a subsample for F, calcium, zinc and iron; urine samples will be measured for F, calcium and creatinine (to correct spot urine). Hemoglobin will be measured as an indicator of overall nutritional status in women and children. Nutritional status of young children (6-18 mo) and of their mothers prior and after the intervention (by 6 months) will be assessed. between 6 and 12 month there will be monitoring for sustainability of chilckens in the community; for continued use of egg (in children) and ESP (in women); during this time the control group will receive chickens and also undergo monitoring. The study will take place in the Rift valley of Southern Ethiopia. Identification of the knowledge, attitude and practices (KAP) of mothers on egg consumption will be done at baseline and at the end ("endline"). Caregivers will be instructed to give each child 1 egg (cooked) per day in the intervention, and one "bottle cap" of eggshell powder (1000 mg calcium) per day for themselves. Families receiving chickens will be instructed on cage construction. Throughout the study, any problems arising in keeping chickens will be recorded in order to assess the feasibility and practicality of raising chickens as way to mitigate fluorosis and improve nutritional status.

DETAILED DESCRIPTION:
This is a Proof of Principle study with a treatment ("Intervention") group and a parallel control group for delivering eggshell powder to mothers in the setting of a chilken intervention. The control and intervention groups will come from the same region in southern Ethiopia where fluorosis is known to occur, with active intervention for 6 months followed by observation for a further 6 months. The Intervention is providing daily eggshell calcium to a subset of mothers, with all eligible young children receiving at least one egg a day. The treatment group consists of mothers and young children in a community where study families will receive two chickens each, and the control group are mothers and young children not having chickens for the first six months, but who will be gifted with chickens at 6 months. Along with receiving chickens, the intervention group will receive training in use of egg, as well as assistance in caring for chickens, throughout the first 6 months. In the second 6-months, the participants' use of eggs will be monitored. In the control group, provision of chickens after 6 months will be accompanied by training but for a shorter duration, and monitoring of use of egg will provide information on whether minimal support can effectively allow for adoption of new food sources into a community.

Study participants are all mothers with children aged between 6-18 months old in two participating kebeles (villages), one randomly assigned as intervention, the other as control. The age group of the child is selected because it is the time of introduction of complementary food and it will be easier to see the clear effect of egg on the children's growth. Mothers are lactating therefore at a time for maximal calcium utilization. While eggs are not commonly eaten in rural Ethiopia, it is due to expense, not to unfamiliarity. In the Intervention community prior to baseline measurements, each family of the mother-child pair will receive two chickens at a "ceremony" that marks the responsibility given to the family to provide one egg per day to the child. In a subset of mothers, they will consent to use eggshell. This is modified from what the investigators did in a pilot study (NCT02791100) and the investigators found use of egg by the child was 85% throughout the 6 month time-period. One lesson learned was to purchase older chickens that are immediately capable of laying eggs. Second, in this intervention the child will not receive ESP.

There will be formal follow-up observation at one community site with focus group discussion and key informant interviews, as a way to assess feasibility and practically of chicken donation in the future. This will be a convenience sample representing participant parents, community leaders, Agriculture Extension workers, Health extension workers, persons who were not directly involved. Those targeted for interviews will be the extension workers from whom feedback will be provided, while focus groups will be held with others who are able to attend a focus group session.

Data checks will be provided by two doctoral students working on the project. Local supervisors will provide guidance. The students have written specific operating procedures (SOP) for all procedures. Missing data will be accounted for, but as this is a community based study group means will be used for most outcome measurements. Comparing of two means/the differences of means between the intervention and control groups will be done using independent two sample t-test. Continuous outcomes will be analyzed using paired t-test. Bivariate analysis will be used to see the overall effect of independent variables and then further multivariate analysis (multiple linear regressions) will be done to see the effect of each independent variable. Both crude and adjusted risk ratio with 95% confidence interval will be reported. Other variables and relevant findings will be also analyzed using proper statistical test/analysis techniques and reported accordingly. P-value of less than 0.05 will be taken as significant

ELIGIBILITY:
Inclusion Criteria:

* All women with a child age 6 to 18 months and their child living permanently in the village
* the woman does not have to be biological mother Exclusion Criteria:
* Exclude families with a child who is known to be allergic to egg
* Exclude families with a child who is diagnosed as malnourished (moderate malnutrition (MAM) or severe malnutrition (SAM)
* Exclude women who do not live with the child

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Children will be male and female but "mothers" will only be female.
Enrollment: 270 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Apparent fluoride absorption | 6 months
  Change in urinary fluoride corrected for creatinine as a measure of F absorption

SECONDARY OUTCOMES:
Growth in young children | 6 months and 12 months
  weight for age
Functional indicators of fluorosis | 6 months
  Physical signs of fluorosis are assessment using a standard questionnaire developed by the investigators and subsequently published (Kebede et al., 2016). Briefly this consists of a questionnaire of signs and symptoms which can be added to obtain a score
Hemoglobin (Hb) | 6 months and 12 months
  Blood levels of Hb
Knowledge, attitude and practices (KAP) for egg | 6 and 12 months
  Questionnaire assessment of KAP
Linear growth in young children | 6 months and 12 months
  length for age

OTHER OUTCOMES:
Inhibition of zinc absorption | 6 months
  serum zinc

CONTACTS AND LOCATIONS:
Overall Officials: Susan Whiting, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Hawassa University, Awasa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
We would find it difficult to keep records for extraction of participant data as the local language will be used to store records.

REFERENCES:
- [Background] Kebede A, N Retta, C Abuye, SJ Whiting, M Kassaw, T Zeru, MW Yohannes, D Zerfu, M Tessema, MK. Malde. Minimizing bioavailability of fluoride through addition of calcium-magnesium citrate or a calcium and magnesium-containing vegetable to the diets of growing rats. International Journal of Biochemistry Research & Review. 10(2): 1-8. 2016a
- [Background] Kebede A, Retta N, Abuye C, Whiting SJ, Kassaw M, Zeru T, Tessema M, Kjellevold M. Dietary Fluoride Intake and Associated Skeletal and Dental Fluorosis in School Age Children in Rural Ethiopian Rift Valley. Int J Environ Res Public Health. 2016 Jul 26;13(8):756. doi: 10.3390/ijerph13080756. PMID 27472351
- [Derived] Mulualem D, Hailu D, Tessema M, Whiting SJ. Efficacy of Calcium-Containing Eggshell Powder Supplementation on Urinary Fluoride and Fluorosis Symptoms in Women in the Ethiopian Rift Valley. Nutrients. 2021 Mar 24;13(4):1052. doi: 10.3390/nu13041052. PMID 33804976